CLINICAL TRIAL: NCT02432079
Title: Molecular Genetics of Heterotaxy and Related Congenital Heart Defects
Status: Recruiting | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Stephanie Ware, Professor of Pediatrics and Medical and Molecular Genetics, Indiana University
Other Study IDs: 1403871897
Record Dates: First submitted 2015-04-28; First posted 2015-05-01 (Estimated); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Heterotaxy Syndrome; Congenital Heart Defects
Keywords: Abnormalities, Multiple; Asplenia; Bilary Atresia; Birth Defect; Cardiovascular Abnormalities; Cardiovascular Diseases; Congenital Abnormalities; Congenital Heart Disease; Dextrocardia Syndrome; Disturbed Internal Organ Positioning; Genetics; Genetic Testing; Heart Defects, Congenital; Heart Diseases; Heterotaxy syndrome; Intestinal malrotation; Laterality; Left Atrial Isomerism; Pediatrics; Polysplenia; Right Atrial Isomerism; Splenic Diseases; Cilia; Situs inversus; Dextrocardia
MeSH Terms: conditions — Heterotaxy Syndrome; Heart Defects, Congenital; Abnormalities, Multiple; Congenital Abnormalities; Cardiovascular Abnormalities; Cardiovascular Diseases; Heart Diseases; Volvulus Of Midgut; Splenic Diseases; Situs Inversus; Dextrocardia

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood, Tissue Sample, Cheek Swabs, Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heterotaxy and congenital heart defects: Patients and family members with heterotaxy and related congenital heart defects

SUMMARY:
The goal of this study is to obtain specimens and data from individuals and their families with heterotaxy and related congenital heart defects in order to clarify the molecular genetics of this disorder. The knowledge gained from the analysis of this information will provide the basis for future genetic counseling as well as contribute to knowledge about the biology of normal and abnormal development of left-right anatomic asymmetry.

DETAILED DESCRIPTION:
Heterotaxy syndrome is a rare birth defect that involves the heart and other organs. Many cases are genetic. Fundamental lack of information about the genetic basis of heterotaxy and related congenital heart defects in the vast majority of children has hindered management and therapy. The study outlined in this protocol is designed to obtain information about the causes of heterotaxy and related congenital heart defects. In this study, investigators will perform genetic analyses on patients with heterotaxy and related congenital heart defects, or individuals at risk for these abnormalities. The investigators will collect medical information related to symptoms and disease course. These results will provide important information on the causes, management, and prognosis of heterotaxy and related congenital heart defects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with heterotaxy and related congenital heart defects
* Family members of subjects with heterotaxy and related congenital heart defects

Exclusion Criteria:

* Subjects without heterotaxy and related congenital heart defects
* Family members of subjects without heterotaxy and related congenital heart defects

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: children affected with heterotaxy syndrome and/or congenital heart defects and their relatives
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2009-07; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Clarify Molecular Genetics of Heterotaxy and Related Congenital Heart Defects | 8 years
  These results will provide important information on the causes, management, and prognosis of heterotaxy and related congenital heart defects. This will provide the basis for future genetic testing and genetic counseling as well as contribute to knowledge about the biology of normal and abnormal development of left-right asymmetry.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie M. Ware, MD, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States